CLINICAL TRIAL: NCT01775657
Title: Digital Versus Analog Pleural Drainage Following Pulmonary Resection
Acronym: DiVA Phase II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20120228-01H
Record Dates: First submitted 2012-11-29; First posted 2013-01-25 (Estimated); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Air Leak; Lobectomy; Wedge Resection; Segmentectomy
Keywords: pulmonary air leak; Thopaz; digital; analog; randomized

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Air leak present - Analogue (Experimental): Patients randomized to Pleur Evac (Analogue drainage) monitoring system, air leak present.
  Interventions: Device: Pleur Evac (Analogue drainage)
- Air leak absent - Analogue (Pleur Evac) (Active Comparator): Patients randomized to Pleur Evac (Analogue drainage) monitoring system, no air leak present
  Interventions: Device: Pleur Evac (Analogue drainage)
- Air leak present - Digital (Thopaz) (Experimental): Patients with an air leak present, randomized to Thopaz (digital drainage) monitoring system.
  Interventions: Device: Thopaz (Digital drainage)
- Air leak absent - Digital (Thopaz) (Active Comparator): Patients randomized to digital system, no air leak present.
  Interventions: Device: Thopaz (Digital drainage)

INTERVENTIONS:
Device: Thopaz (Digital drainage)
  Other Names: Thopaz, Medela Switzerland
  Arms: Air leak absent - Digital (Thopaz); Air leak present - Digital (Thopaz)
Device: Pleur Evac (Analogue drainage)
  Other Names: Pleur Evac A-6002-08, Teleflex Inc, Research Triangle Park, NC, USA
  Arms: Air leak absent - Analogue (Pleur Evac); Air leak present - Analogue

SUMMARY:
This study will evaluate the impact of continuous, digital pulmonary air leak monitoring on the duration of pleural drainage after lung resection in patients with and without a pulmonary air leak on postoperative day 1.

Patients undergoing pulmonary resection who fit the inclusion criteria will be identified pre-operatively. Patients within two groups (air leak and no air leak) will be randomized to receive either the analogue system or the digital system. Both systems are approved for use in hospitals by Health Canada. There will be 88 patients in each air leak group.

Hypothesis: Continuous, quantitative monitoring of PAL following lung resection leads to an improvement in primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

Elective pulmonary resection (i.e. wedge, segmentectomy, lobectomy, bilobectomy) for benign or neoplastic disease

Exclusion Criteria:

1. Development of tension pneumothorax
2. Pneumonectomy
3. Patient no longer within planned randomization window
4. Plan to remove or removal of all chest drains within 36 hours of surgery
5. Inability to provide informed consent
6. Age < 18 years
7. Patient was previously randomized following pulmonary resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Overall length of hospitalization | Up to 5 days post-op (average)

SECONDARY OUTCOMES:
Time to first pleural drain removal | Over 24 hours post-op

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Gilbert, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital, General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gilbert S, McGuire AL, Maghera S, Sundaresan SR, Seely AJ, Maziak DE, Shamji FM, Villeneuve PJ. Randomized trial of digital versus analog pleural drainage in patients with or without a pulmonary air leak after lung resection. J Thorac Cardiovasc Surg. 2015 Nov;150(5):1243-9. doi: 10.1016/j.jtcvs.2015.08.051. Epub 2015 Aug 28. PMID 26409729